CLINICAL TRIAL: NCT00771420
Title: A Double-blind, Placebo-controlled, Single Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CAM-3001 in Patients With Rheumatoid Arthritis.
Brief Title: A Single Dose Study of the CAM-3001 in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune Ltd (Industry)
Responsible Party: Sponsor
Organization: MedImmune LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAM-3001-0702
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — mavrilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1 (Active Comparator): 0.01mg/kg and 0.03mg/kg CAM-3001
  Interventions: Drug: CAM-3001
- 2 (Active Comparator): 0.1mg/kg CAM-3001
  Interventions: Drug: CAM-3001
- 3 (Active Comparator): 0.3mg/kg CAM-3001
  Interventions: Drug: CAM-3001
- 4 (Active Comparator): 1.0mg/kg CAM-3001
  Interventions: Drug: CAM-3001
- 5 (Active Comparator): 3.0mg/kgCAM-3001
  Interventions: Drug: CAM-3001
- 6 (Active Comparator): 10.0mg/kg CAM-3001
  Interventions: Drug: CAM-3001
- 7 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CAM-3001 — A single patient shall be dosed with a dose of 0.01mg/kg of CAM-3001 followed no sooner than 24 hours later by a second patient at a dose of 0.03mg/kg.
  Other Names: Mavrilimumab
  Arms: 1
Drug: CAM-3001 — Dosed at 0.1mg/kg.
  Other Names: Mavrilimumab
  Arms: 2
Drug: CAM-3001 — Dosed at 0.3mg/kg
  Other Names: Mavrilimumab
  Arms: 3
Drug: CAM-3001 — Dosed at 1.0 mg/kg.
  Other Names: Mavrilimumab
  Arms: 4
Drug: CAM-3001 — Dosed at 3.0 mg/kg.
  Other Names: Mavriliumab
  Arms: 5
Drug: CAM-3001 — Dosed at 10 mg/kg.
  Other Names: Mavrilimumab
  Arms: 6
Other: Placebo — Active: Placebo 5:1 for arms 2-6
  Arms: 7

SUMMARY:
Investigate safety and tolerability of the escalating dose of CAM-3001 in patients.

DETAILED DESCRIPTION:
To investigate the safety and tolerability of escalating single doses of CAM-3001 in patients with RA; To investigate the pharmacokinetics of single doses of CAM-3001 in RA patients; To investigate the pharmacodynamics of single doses of CAM-3001 in RA patients; To investigate the preliminary clinical effects of CAM-3001 on the signs and symptoms of RA.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent, prior to any study related procedures
* Male and female patients aged 18-70 years at the screening visit
* Use of an appropriate method of contraception
* A diagnosis of adult onset rheumatoid arthritis of at least 6 months duration as defined by the 1987 ACR classification criteria - ACR functional class I, II or III
* Treatment with methotrexate for at least 3 months and stable dose 10mg - 25mg / week for ≥ 8 weeks prior to the baseline visit
* Availability of clear chest X-ray (i.e. no evidence of TB, chest infection or cardiac failure). Patients who are clinically asymptomatic with minor changes consistent with rheumatoid lung are acceptable.
* Stable mild or inactive rheumatoid arthritis where in the opinion of the investigator it is unlikely that a change in the patient's therapeutic regimen would be required during the subsequent 3 months.
* DAS28 ≤ 4.8 for at least 3 months prior to the baseline visit

Exclusion Criteria:

* Relating to RA
* Diagnosis of any other inflammatory arthritis (e.g. psoriatic arthritis or ankylosing spondylitis), or a diagnosis of a secondary, non-inflammatory type of arthritis (e.g. osteoarthritis or fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with the evaluation of the effect of CAM-3001 on the patient's primary diagnosis of rheumatoid arthritis Relating to Previous Clinical Trials and Biologic Therapies
* Administration of any investigational or experimental non-biologic therapy in the 12 weeks prior to the baseline visit
* Administration of any biologic therapy within 6 months prior to the baseline visit Relating to Concomitant Medications
* Use of prohibited concomitant medications, which might confound the interpretation of the study data Relating to Medical History
* Female patients who are pregnant or breast-feeding, or who plan to become pregnant during the trial or during the 24 weeks after administration of CAM-3001
* Male or female patients not willing to use reliable methods of birth control for the duration of the study
* A history of TB, or clinical/radiographic evidence of TB, or positive TB test
* A history or current symptoms and signs of chronic infection, or recent (within 6 months prior to screening visit) serious infection including herpes zoster
* Patients at a high risk of infection e.g. a history of an infected joint prosthesis at any time with that prosthesis still in situ, leg ulcers, indwelling urinary catheter, persistent or recurrent chest infections
* Neutrophil count < 1000 x 106 cells/L
* A positive hepatitis B surface antigen test and/or hepatitis C antibody test result
* A positive test for human immunodeficiency virus (HIV) infection
* Receipt of live (attenuated) vaccine within the 4 weeks prior to baseline or during the study
* Current or recent history of significant renal, hepatic, haematological, immunological (other than RA), gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease which would interfere with the patient's participation in the trial. Patients with mild and stable asthma or mild and stable Chronic Obstructive Pulmonary Disease (COPD) may be included at the discretion of the Investigator
* Active malignancy or lymphoproliferative disorder of any type, or a history of malignancy except for basal cell carcinoma of the skin that has been excised prior to the screening visit
* Suspected alcohol or substance abuse
* Donation of ≥ 400mL of blood within 8 weeks prior to baseline
* Any other significant medical condition which in the opinion of the investigator might increase the risk to the patient or confound the interpretation of the data
* Individuals who are legally institutionalised

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events • Changes in vital signs, ECG, lung function tests and clinical laboratory values | End of study

SECONDARY OUTCOMES:
Pharmacokinetic parameters of CAM-3001 will be calculated and tabulated descriptively for each dose group: | Day 28 post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Ehsanollah Esfandiari, PhD MD, Study Director — MedImmune LLC
Locations (1):
- Charite Research Organization GmbH, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Burmester GR, Feist E, Sleeman MA, Wang B, White B, Magrini F. Mavrilimumab, a human monoclonal antibody targeting GM-CSF receptor-alpha, in subjects with rheumatoid arthritis: a randomised, double-blind, placebo-controlled, phase I, first-in-human study. Ann Rheum Dis. 2011 Sep;70(9):1542-9. doi: 10.1136/ard.2010.146225. Epub 2011 May 25. PMID 21613310